CLINICAL TRIAL: NCT07045844
Title: The Effects of Different Enteral Feeding Regimens on Necrotizing Enterocolitis, Mortality, and Neurodevelopment in Very Preterm Infants: A Multicenter Double-Randomized Trial
Brief Title: Effects of Enteral Feeding Regimens on NEC, Mortality, and Neurodevelopment in Very Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Yanping Xu, Dr., The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-IRB-0232-P-02
Record Dates: First submitted 2025-06-17; First posted 2025-07-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Very Preterm Infant; Necrotizing Enterocolitis (NEC)
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pasteurized Donor Milk for Insufficient Breastfeeding (Experimental): Participants receive pasteurized donor human milk (pHDM) as supplemental feeding when the clinician determines maternal milk supply is insufficient.
  Interventions: Dietary Supplement: Pasteurized Donor Milk for Insufficient Breastfeeding; Dietary Supplement: Routine fortification; Dietary Supplement: Rescue fortification
- Preterm formula for Insufficient Breastfeeding (Experimental): Participants receive preterm formula (PTF) as supplemental feeding when the clinician determines maternal milk supply is insufficient.
  Interventions: Dietary Supplement: Preterm Formula for Insufficient Breastfeeding; Dietary Supplement: Routine fortification; Dietary Supplement: Rescue fortification

INTERVENTIONS:
Dietary Supplement: Pasteurized Donor Milk for Insufficient Breastfeeding — Participants receive pasteurized donor human milk (pHDM) as supplemental feeding when the clinician determines maternal milk supply is insufficient.
  Randomization 1 will occur when the clinician determines that supplemental feeding is required due to insufficient breast milk supply.
  Arms: Pasteurized Donor Milk for Insufficient Breastfeeding
Dietary Supplement: Preterm Formula for Insufficient Breastfeeding — Participants receive preterm formula (PTF) as supplemental feeding when the clinician determines maternal milk supply is insufficient.
  Randomization 1 will occur when the clinician determines that supplemental feeding is required due to insufficient breast milk supply.
  Arms: Preterm formula for Insufficient Breastfeeding
Dietary Supplement: Routine fortification — Randomization 2 will be conducted when the total daily intake of human milk (including own mother's milk [OMM] and/or donor pasteurized human milk [pHDM] ) reaches between 60-120 mL/kg
Dietary Supplement: Rescue fortification — Randomization 2 will be conducted: Add fortifiers when the infant meets predefined criteria for growth faltering (Preterm infants exhibit a sustained decline in growth velocity for weight, length, or head circumference, demonstrated by a downward crossing of centiles on growth curves, despite tolerating and consuming at least 180 mL/kg/day of breast milk or formula. Blood urea levels in these infants remain consistently below 1.5 mmol/L, and there are no severe complications such as active sepsis or the need for vasoactive medications to maintain circulatory stability. Chronic sodium depletion has also been ruled out, as this condition alone can lead to growth failure. Additionally, preterm infants are unable to tolerate high-volume feeding of 180 mL/kg/day due to specific reasons, such as severe gastroesophageal reflux or the presence of a high-output stoma following surgical procedures).

SUMMARY:
The goal of this clinical trial is to evaluate whether supplementing with pasteurized donor human milk (pHDM) or preterm formula (PTF) when own mother's milk (OMM) is insufficient can improve outcomes in very preterm infants born before 29 weeks of gestation. It also aims to assess whether routine use of human milk fortifiers benefits this population. The main questions it aims to answer are:

Does supplementing OMM with pHDM or PTF improve survival without surgery-requiring necrotizing enterocolitis (NEC) by 34 weeks corrected gestational age? Is routine fortification of human milk better than selective fortification based on growth faltering?

Researchers will compare:

pHDM vs. PTF to see which better supports survival without severe NEC. Routine fortification vs. selective fortification to assess the impact on growth and long-term neurodevelopment.

Participants will:

Be randomized twice:

* First, within the first week of life to receive either pHDM or PTF when OMM is insufficient
* Second, in the second week of life to receive either routine fortification or selective fortification only if growth faltering occurs Receive feeding and care as per standard clinical practice Complete neurodevelopmental assessment at 2 years corrected age using the PARCA-R tool (no additional study visits required) This multicenter, double-randomized, open-label randomized controlled trial is embedded in routine neonatal care and uses real-world data to assess both short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth less than 29 weeks;
* No contraindications to enteral feeding;
* Mother is willing to breastfeed.

Exclusion Criteria:

* For Randomization Group 1: If the infant has already received pasteurized human donor milk (pHDM), preterm formula (PTF), or nutritional fortifiers;
* For Randomization Group 2: If the infant is exclusively fed with preterm formula and the mother has no intention to express breast milk;

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2324 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Survival without surgical NEC | 34 weeks corrected gestational age
  Survival to 34 weeks corrected gestational age without surgical necrotizing enterocolitis (NEC)

SECONDARY OUTCOMES:
NEC requiring surgical intervention | 34 weeks gestational age
Survival | 28 days after birth
Survival that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Survival: Survival outcome indicators measure the success of enduring life-threatening conditions, eg. survival rate.
Medically treated NEC that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Medically treated NEC: Diagnosis of necrotizing enterocolitis that required medical (non-surgical) treatment, such as bowel rest and antibiotic therapy.
Treated retinopathy of prematurity (ROP) that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Treated retinopathy of prematurity (ROP): ROP that progressed to a stage requiring medical or surgical intervention, including laser therapy or intravitreal injections.
Hearing impairment that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Hearing impairment: Documented hearing loss identified through newborn hearing screening or diagnostic audiology tests, potentially requiring follow-up or intervention.
Severe brain injury that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Severe brain injury: Presence of significant brain injury such as Grade III or IV intraventricular hemorrhage (IVH) or periventricular leukomalacia (PVL) as diagnosed by cranial imaging.
Length of hospital stay | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Length of hospital stay: Total number of days from birth until discharge from the hospital.
Number of episodes of bloodstream infection that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Number of episodes of bloodstream infection: Total number of confirmed bloodstream infections (positive blood cultures) during the hospital stay.
Events that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Number of days of antibiotic treatment: Cumulative number of days the infant received systemic antibiotic therapy during hospitalization.
Number of days on parenteral nutrition that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Number of days on parenteral nutrition: Total number of days the infant received intravenous nutritional support due to inability to tolerate full enteral feeds.
Number of days of NPO that occurred during hospitalization | From birth until hospital discharge (up to approximately 44 weeks postmenstrual age)
  Number of days of NPO: Total number of days the infant was designated "nil per os" (NPO), meaning no enteral feeding was given.
Body weight | From birth until 2 years corrected age.
  Growth parameters (weight): Measurements of the infant's body weight at 2 years corrected age.
Body length | From birth until 2 years corrected age.
  Body length: Measurements of the infant's body length at 2 years corrected age.
Head circumference | From birth until 2 years corrected age.
  Head circumference: Measurements of the infant's head circumference at 2 years corrected age.
Parent Report of Children's Abilities-Revised (PARCA-R) assessment | At 2 years corrected age
  Survival without moderate to severe cognitive or language impairment. PARCA-R stands for Parent Report of Children's Abilities-Revised. It is a parent completed questionnaire that can be used to assess children's cognitive and language development at 24 months of age.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Yongkang Maternity and Child Health Care Hospital, Guli, Zhejiang
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Women's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hangzhou Women's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jiaxing Maternity and Child Health Care Hospital, Jiaxing, Zhejiang
  - Ningbo Women and Children's Hospital (The Affiliated Women and Children's Hospital of Ningbo University), Ningbo, Zhejiang
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Yiwu Maternity and Child Health Care Hospital (Yiwu Branch of The Children's Hospital, Zhejiang University School of Medicine), Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT07045844/Prot_SAP_ICF_001.pdf